CLINICAL TRIAL: NCT03461341
Title: ENSURE: European iNvestigation of SUrveillance After Resection for Esophageal Cancer
Brief Title: European iNvestigation of SUrveillance After Resection for Esophageal Cancer
Acronym: ENSURE
Status: Completed | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: St Mary's Hospital, Paddington, London (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Other Study IDs: SJHDOS201801
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Cancer; Metastatic Cancer; Recurrent Esophageal Cancer; Chemoradiation; Chemotherapy; Radiation; Surgery
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients post curative intent surgery for esophageal cancer: Patients post potentially curative surgery for cTxNxM0 esophageal or esophagogastric junction (Siewert type I, II and III) cancer.
  Interventions: Other: High intensity postoperative oncologic surveillance

INTERVENTIONS:
Other: High intensity postoperative oncologic surveillance — High intensity surveillance protocol using routine cross-sectional imaging (computed tomography or positron emission tomography with computed tomography).
  Other Names: Screening for recurrence; Oncologic surveillance; Imaging follow-up

SUMMARY:
The ENSURE study will comprise two phases.

Phase 1: European multicenter survey of surveillance protocols after esophageal cancer surgery

ENSURE questionnaire will be circulated to representatives from participating European countries.

Phase 2: European multicenter retrospective observational study of the impact of postoperative surveillance protocols on oncologic outcome and HR-QL

Phase 2 will constitute a retrospective observational study of patients undergoing treatment with curative intent for esophageal cancer at participating Centers from June 2009 to June 2015.

DETAILED DESCRIPTION:
Despite significant improvements in oncologic outcome for patients with esophageal cancer, with increased early detection and greater utilization of multimodal protocols,approximately 50% and 20% patients with locally advanced and localized disease treated with curative intent will develop disease recurrence within 5 years. After completion of treatment, there is little evidence to guide surveillance strategies, and whether routine clinical, biochemical, radiologic or endoscopic follow-up is associated with improved oncologic outcomes, or health-related quality of life (HR-QL), is unknown. This is in contrast to colorectal cancer, where meta-analyses demonstrate a significant overall survival (OS) benefit among patients undergoing intensive surveillance, likely driven by a proportion of patients achieving long-term survival following salvage treatments for oligometastatic disease. Importantly, intensive surveillance in colorectal cancer did not adversely impact HR-QL in survivorship.

In esophageal cancer, a lack of quality to indicate that aggressive treatment of recurrent disease provided an OS benefit had previously limited the rationale for intensive oncologic surveillance in this cohort. However, increasingly reports of long-term survival after salvage surgery for recurrent esophageal cancer among patients treated with esophagectomy as a component of initial treatment are emerging. For example, Depypere et al. reported that among the 15% of patients with isolated local recurrence or single solid organ metastasis who were treated surgically, 5-year survival from time of recurrence was 50% (median 55 months). This is in keeping with data from Schipper et al. who report 44% and 35% 3- and 5-year survival, respectively, in the minority of patients for whom R0 re-resection of local recurrence was possible. Furthermore, while meta-analysis now confirms the survival benefit of palliative chemotherapy (HR 0.81, 95% CI 0.71 to 0.92), and targeted therapy (HR 0.75, 95% CI 0.68 to 0.84), the independent impact of timing of intervention, and disease volume, on OS in the setting of recurrent disease is unclear.

Indeed, no randomized controlled trial has compared oncologic outcomes among cohorts undergoing different surveillance protocols, and only two retrospective observational studies have directly addressed this question. In a study from Canada, Peixoto et al. compared survival outcomes among 292 patients with gastroesophageal cancers (58% esophageal and junctional, with 23% treated with definitive chemoradiation only), undergoing four different surveillance modalities (discharge to General Practitioner, or Medical Oncology follow-up with either clinical, clinical and biochemical, or clinical and radiologic/endoscopic surveillance). There was no difference in recurrence-free or OS according to surveillance strategy on univariable or multivariable analysis. However, recent data from Sisic et al. advise caution in interpretation of the former study. Among 587 patients undergoing either high intensity radiologic or standard clinical surveillance after potentially curative treatment for gastric (47%) or junctional (53%) adenocarcinoma, intensive surveillance independently predicted OS on multivariable analysis and was associated with an approximate 5% increase in OS at 3 and 5 years. Notably, among patients who developed disease recurrence, OS was significantly greater (median 40 versus 19 months) for those with radiologically-detected versus clinical recurrence, and for those who underwent metastectomy (n = 29, 5% of total population) versus other treatments (median 66 versus 25 months), similar to previous series. Although this likely reflects, at least in part, inherent differences in disease biology and volume among those who recur symptomatically versus radiologically, patients undergoing high intensity surveillance were more likely to have treatment for recurrence, with a proportion of these achieving long-term survival (n = 11, 2% of total population). Though limited, these data indicate that intensive surveillance may provide benefit for the small proportion of patients who may be treated with curative intent for low volume recurrence.

Given the limited evidence to support postoperative surveillance protocols in esophageal cancer, it is unsurprising that international guidelines also fail to reach consensus on this topic. For example, the National Comprehensive Cancer Network (NCCN) recommend regular cross-sectional imaging with computed tomography (CT) for all patients with locally advanced disease (cT2-4 Nany) post multimodal therapy, and consideration of regular surveillance CT among patients with T1b Nany treated with upfront esophagectomy, up to 3 years postoperatively, with endoscopic surveillance only in the case of residual Barrett's esophagus. In contrast, European Society for Medical Oncology (ESMO) guidelines highlight a lack of evidence to support the role of postoperative surveillance protocols to improve oncologic outcomes, and determine that follow-up should concentrate on symptoms, nutrition and psychological support, and neither routine imaging nor endoscopic surveillance is advocated.

As indicated in the ESMO and ASGBI surveillance recommendations, there are potential additional benefits to postoperative surveillance protocols. Routine clinical surveillance may facilitate identification and management of late post treatment morbidity such as anastomotic stricture, post thoracotomy pain, malabsorption, altered appetite and dumping syndrome. Furthermore, data from the Netherlands indicate that patients exhibit a strong preference for routine imaging surveillance after esophagectomy, with 67% preferring imaging even if this approach would not provide a survival benefit.19 This is in keeping with UK colorectal cancer data demonstrating that although surveillance is associated with transient anxiety, negative test results provide significant reassurance for the majority. Interestingly, similar to the Dutch data, most patients (78%) stated that they would value finding out about the presence of recurrence, even if there would be no survival benefit. This would provide evidence to counter the concern that postoperative surveillance may negatively influence HR-QL, either through increased anxiety related to surveillance investigations, or earlier diagnosis of otherwise asymptomatic patients with recurrent disease.

Examining surveillance practices internationally, there is significant variability in the utilization of biochemical, radiologic and endoscopic surveillance. In Japan, a nationwide survey found that high intensity surveillance was common, and notably endoscopic surveillance was frequently utilized (85%), in contrast to Australia and New Zealand where only 6% of surgeons opted to undertake routine endoscopic surveillance of asymptomatic patients after potentially curative esophagectomy. The European Registration of Cancer Care (EURECCA) Upper Gastrointestinal group included a brief summary of postoperative surveillance protocols for esophagogastric adenocarcinoma among the 10 participating Centers in a recent publication on clinical pathways. Importantly, this demonstrated clear differences across European Centers in key elements of surveillance, such as the routine use of CT (in 40%) and tumor markers (in 40%), but did not describe endoscopic surveillance protocols or duration of surveillance, while oncologic outcomes according to surveillance intensity were not assessed.

Given these major differences in surveillance intensity and modality across Europe, with otherwise similar population demographics and treatment pathways, we in Europe are uniquely poised to further study the impact of surveillance with respect to oncologic outcome, and HR-QL, after potentially curative surgery for esophageal cancer. Therefore, the primary aims of this European collaborative multicenter study are:

1. Firstly, to characterize differences in postoperative oncologic surveillance protocols across European esophageal cancer centers, and
2. To determine the independent impact of high intensity surveillance (HIS) on disease-specific and overall survival.

ELIGIBILITY:
Inclusion criteria

1. Age 18 years and above
2. Underwent surgery with curative intent for cTxNxM0 esophageal or esophagogastric junction (Siewert type I, II and III) cancer
3. Salvage surgery after failure of primary endoscopic or oncologic treatment will be included

Exclusion criteria

1. Endoscopic therapy or definitive oncological treatment as sole therapy for esophageal cancer
2. Missing follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 2 will constitute a retrospective observational study of patients undergoing treatment with curative intent for esophageal cancer at participating Centers from June 2009 to June 2015.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-06-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (months) | Minimum 3 year follow-up for all patients
  Overall survival in months will be compared by Kaplan-Meier methods and using multivariable Cox proportional hazards regression, adjusting for known prognostic factors, to determine the independent impact of high intensity surveillance on survival outcome.
Disease-specific survival (months) | Minimum 3 year follow-up for all patients
  Disease-specific survival in months will be compared by Kaplan-Meier methods and using multivariable Cox proportional hazards regression, adjusting for known prognostic factors, to determine the independent impact of high intensity surveillance on survival outcome.
Utilisation of routine surveillance imaging across European Centers | 2009 - 2015
  The proportion of European Centers utilising routine postperative oncologic surveillance imaging will be determined by email survey.

SECONDARY OUTCOMES:
Isolated solid organ metastasis (ISOM) at first recurrence | Minimum 3 year follow-up for all patients
  Proportion of patients in high intensity versus standard surveillance groups with ISOM at first recurrence.
Isolated local recurrence (ILR) at first recurrence | Minimum 3 year follow-up for all patients
  Proportion of patients in high intensity versus standard surveillance groups with ILR at first recurrence.
Health-related quality of life (HR-QL) as assessed by EORTC QLQ-C30 questionnaire | At one year postoperatively
  "Overall health" score among disease-free patients at least one year postoperatively compared between high intensity and standard surveillance groups.

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MD FRCS, Principal Investigator — St. James's Hospital, Dublin, Ireland; George B Hanna, PhD FRCS, Principal Investigator — St. Mary's Hospital, London, United Kingdom; Magnus Nilsson, MD FRCS, Principal Investigator — Karolinska Institutet
Locations (3):
- Department of Surgery, St. James's Hospital, Dublin, Ireland
- Karolinska Institutet, Stockholm, Sweden
- Department of Surgery and Cancer, 10th Floor, QEQM building, St. Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antonowicz SS, Lorenzi B, Parker M, Tang CB, Harvey M, Kadirkamanathan SS. Annual computed tomography scans do not improve outcomes following esophagectomy for cancer: a 10-year UK experience. Dis Esophagus. 2015 May-Jun;28(4):365-70. doi: 10.1111/dote.12209. Epub 2014 Mar 20. PMID 24649807
- [Background] Messager M, de Steur W, Boelens PG, Jensen LS, Mariette C, Reynolds JV, Osorio J, Pera M, Johansson J, Kolodziejczyk P, Roviello F, De Manzoni G, Monig SP, Allum WH; EURECCA Upper GI group (European Registration of Cancer Care). Description and analysis of clinical pathways for oesophago-gastric adenocarcinoma, in 10 European countries (the EURECCA upper gastro intestinal group - European Registration of Cancer Care). Eur J Surg Oncol. 2016 Sep;42(9):1432-47. doi: 10.1016/j.ejso.2016.01.001. Epub 2016 Feb 6. PMID 26898839
- [Background] Peixoto RD, Lim HJ, Kim H, Abdullah A, Cheung WY. Patterns of surveillance following curative intent therapy for gastroesophageal cancer. J Gastrointest Cancer. 2014 Sep;45(3):325-33. doi: 10.1007/s12029-014-9601-3. PMID 24756830
- [Background] Depypere L, Lerut T, Moons J, Coosemans W, Decker G, Van Veer H, De Leyn P, Nafteux P. Isolated local recurrence or solitary solid organ metastasis after esophagectomy for cancer is not the end of the road. Dis Esophagus. 2017 Jan 1;30(1):1-8. doi: 10.1111/dote.12508. PMID 27704661
- [Background] Sisic L, Strowitzki MJ, Blank S, Nienhueser H, Dorr S, Haag GM, Jager D, Ott K, Buchler MW, Ulrich A, Schmidt T. Postoperative follow-up programs improve survival in curatively resected gastric and junctional cancer patients: a propensity score matched analysis. Gastric Cancer. 2018 May;21(3):552-568. doi: 10.1007/s10120-017-0751-4. Epub 2017 Jul 24. PMID 28741059
- [Background] Abate E, DeMeester SR, Zehetner J, Oezcelik A, Ayazi S, Costales J, Banki F, Lipham JC, Hagen JA, DeMeester TR. Recurrence after esophagectomy for adenocarcinoma: defining optimal follow-up intervals and testing. J Am Coll Surg. 2010 Apr;210(4):428-35. doi: 10.1016/j.jamcollsurg.2010.01.006. PMID 20347734
- [Derived] Elliott JA, Markar SR, Klevebro F, Johar A, Goense L, Lagergren P, Zaninotto G, van Hillegersberg R, van Berge Henegouwen MI, Nilsson M, Hanna GB, Reynolds JV; ENSURE Study Group. An International Multicenter Study Exploring Whether Surveillance After Esophageal Cancer Surgery Impacts Oncological and Quality of Life Outcomes (ENSURE). Ann Surg. 2023 May 1;277(5):e1035-e1044. doi: 10.1097/SLA.0000000000005378. Epub 2022 Jan 27. PMID 35129466